CLINICAL TRIAL: NCT06855966
Title: Assessment of End-Tidal Carbon Dioxide Changes in Response to Passive Leg Raise for Guiding Fluid Management in Lung Resections: a Randomized Controlled Trial
Brief Title: Feasibility of ETCO₂ Changes During Passive Leg Raise for Fluid Management in Lung Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Havva Suheyla Akin Uzan, doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC-AR-HSAU-01
Record Dates: First submitted 2025-02-05; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): PLR applied to this group as well as other two groups. An increase of 2mmHg detected in these patients. However, this group received the conventional fluid replacement regimen of the institution of the investigators, which is 2ml/kg/hr crystalloid infusion. The blood pressure is monitorized continually in each patient from a radial artery cannula, and an infusion of noradrenaline started if mean arterial pressure persisted below 65 mmHg.The blood product replacement plan is keeping the hemoglobin level over 10 g/dL for patients with coronary artery disease and 8 g/dL for other patients.
- Study (Experimental): PLR applied to this group as well as other two groups. A 2 mmHg increase at EtCO2 detected at 1st minute of PLR. The patients in this group named as study group and received a 250 ml of crystalloid bolus. These patients also received another 250 ml crystalloid bolus if mean arterial pressure is below 65 mmHg at the end of infusion.The blood pressure is monitorized continually in each patient from a radial artery cannula, and an infusion of noradrenaline started if mean arterial pressure persisted below 65 mmHg after total of 500 ml crystalloid bolus.The blood product replacement plan is keeping the hemoglobin level over 10 g/dL for patients with coronary artery disease and 8 g/dL for other patients.
  Interventions: Other: 250 ml crystalloid bolus infusion
- Unresponsive (No Intervention): Patients in this group showed no change at End tidal carbon dioxide measurement as a response to PLR and received the conventional fluid replacement regimen of the institution of the investigators, which is 2ml/kg/hr crystalloid infusion.The blood pressure is monitorized continually in each patient from a radial artery cannula, and an infusion of noradrenaline started if mean arterial pressure persisted below 65 mmHg.The blood product replacement plan is keeping the hemoglobin level over 10 g/dL for patients with coronary artery disease and 8 g/dL for other patients.

INTERVENTIONS:
Other: 250 ml crystalloid bolus infusion — In thoracic surgical setting, restrictive fluid replacement is widely accepted. However, goal directed fluid therapies can provide a more precise and tailored fluid replacement for each patient. Although ERAS protocols emphasize otherwise, patients still arrive in the operating room with certain deficite, due to prolonged fasting or advanced age. PLR is used as a reversible fluid challenge since the blood which is pooled in the lower extremities as well as splancnic area. End tidal carbon dioxide is monitorized at each patient per American Society of Anesthesia Guideline. In this study, we aimed to assess the feasibility of end tidal carbondioxide changes as a response to passive leg raise maneuer (PLR) for preload optimization in thoracic surgical practice.
  Arms: Study

SUMMARY:
Aim: End tidal carbondioxide pressure (EtCO2) is an indirect indicator of cardiac output (CO) which is monitored in every patient at perioperative setting. The investigators aimed to use increase of EtCO2 as a response to passive leg raising maneuver (PLR) to indicate fluid responsiveness in patients who underwent lung resection with video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
Materials and Methods: 50 patients included who are eligible according to inclusion criteria of the study who underwent lung resection operation via VATS between Agust 2020-March 2021. After a standardized anesthesia induction protocol and intubation, PLR is applied to all patients as soon as anesthesia depth and ventilation stabilized. An increase of 2 mmHg at EtCO2 at first minute of PLR evaluated as "fluid responsive" due to an increase of venous return. Responsive patients divided into two groups as "study" and "control" when unresponsive patiens inclueded into "unresponsive" group. Patients at study group received a fluid bolus (250 ml (and an additional 250 ml if mean arterial pressure remained below 65 mmHg )) in addition to maintainence fluid as control group and unresponsive group received only maintainence fluid. Hemodynamic data, surgery duration, total iv fluid administration, use of blood products, bleeding and urine output during surgery of all patients recorded. Preopretive and postoperative urea, creatinine and lactate levels of all patiens compared. Total iv fluid administration and urine output recorded during postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung resection surgery via VATS
* ASA I-II-III
* Patients older than 18 years

Exclusion Criteria:

* ASA IV or more
* Post operative ICU stay
* Resections greater than lobectomy
* History of renal and heart failure
* Patients younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in End-Tidal Carbon Dioxide (EtCO₂) in Response to Passive Leg Raise (PLR) | Time Frame: Intraoperative (Baseline and 1 Minute After PLR)
  Measurement Method: EtCO₂ (mmHg) will be recorded using a side-stream capnograph integrated into the anesthesia workstation. Baseline EtCO₂ will be measured in the supine position before the PLR maneuver. The PLR maneuver will then be performed by elevating the lower extremities to a 45-degree angle while maintaining a supine upper body position. The position remained for 1 minute and the maximum level of EtCO₂recorded.
  Outcome Definition: A ≥2 mmHg increase in EtCO₂ from baseline within 1 minute of PLR will be classified as a positive response, indicating fluid responsiveness. Patients with an EtCO₂ increase of <2 mmHg will be classified as non-responders.

SECONDARY OUTCOMES:
Change in Serum Urea Levels | Preoperative, 24 hours, and 48 hours postoperatively (if patient remains hospitalized)
  Blood samples will be collected at baseline (preoperative), and at 24 hours postoperatively for all participants. If the patient remains hospitalized at 48 hours, an additional blood sample for urea will be collected. Serum urea (mg/dL) levels will be analyzed using standard laboratory biochemical methods.
Change in Serum Creatinine Levels | Preoperative, 24 hours, and 48 hours postoperatively (if patient remains hospitalized)
  Blood samples will be collected at baseline (preoperative), and at 24 hours postoperatively for all participants. If the patient remains hospitalized at 48 hours, an additional blood sample for creatinine will be collected. Serum creatinine (mg/dL) levels will be analyzed using standard laboratory biochemical methods.
Change in Serum Lactate Levels | Preoperative, 24 hours
  Blood samples will be collected at baseline (preoperative), and at 24 hours postoperatively for all participants. Serum lactate (mmol/L) levels will be analyzed using standard laboratory biochemical methods.

OTHER OUTCOMES:
Correlation Between Pleth Variability Index (PVI) and Fluid Responsiveness Based on EtCO₂ Changes | Time Frame: Intraoperative (Baseline and during 1 Minute of PLR maneuer)
  PVI (%) will be recorded before and after PLR using Masimo Rainbow SET. Correlation between PVI values and EtCO₂-based fluid responsiveness classification (≥2 mmHg EtCO₂ increase) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lale Yuceyar, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa Medical School Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uzan HSA, Yuceyar L, Sayilgan NC. End-tidal CO2 response to passive leg raise for fluid management in lung resections: A randomized controlled trial. Pak J Med Sci. 2025 Dec;41(12):3393-3398. doi: 10.12669/pjms.41.12.12679. PMID 41450995